CLINICAL TRIAL: NCT06211361
Title: Impact of a Cardiac Rehabilitation Program in Patients with Cardiovascular Disease
Brief Title: Cardiac Rehabilitation Program in Patients with Cardiovascular Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Virgen de la Luz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG: 2023/PI0523
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular diseases; heart failure; ischemic heart disease; cardiac rehabilitation; exercise training; cardiopulmonary exercise test; oxygen uptake
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Myocardial Ischemia | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: Our project is a quantitative study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will be included in a cardiac rehabilitation program.
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation — Physical exercise intervention within a cardiac rehabilitation program, lasting 2 months, 3 days per week. The intervention consists of a first part of warm up the large muscle groups, accompanied by breathing exercises, followed by a part of strength and muscular resistance training exercises (upper and lower limbs and abdominal muscles), another part of aerobic exercise part (continuous and interval), using a treadmill or cycle ergometer, and finally a part of stretching exercises and a cool-down phase.
  Other Names: Exercise training program

SUMMARY:
This protocol study aims to evaluate the effectiveness of a cardiac rehabilitation intervention program in patients with cardiovascular diseases to improve both anthropometric and biochemical data, as well as other variables related to cardiovascular disorders (cardiorespiratory fitness, muscle strength, …), and emotional aspects (anxiety, depression).

Additionally, this study aims to evaluate the effectiveness of the cardiac rehabilitation program in improving body composition (waist circumference and body fat percentage), blood pressure and health-related quality of life.

Objectives: i) To assess the functional capacity of patients with a recent cardiovascular event (acute coronary syndrome, onset heart failure, valve or bypass surgery) or with chronic decompensated cardiovascular disease (valvulopathy, pulmonary hypertension, congenital heart disease, heart failure) chronic), ii) to determine the different cardiorespiratory parameters obtained from cardiopulmonary exercise testing (CPET), iii) to determine the lifestyle habits and cardiovascular risk factors, iv) to develop a cardiac rehabilitation program according to and adapted to the need of each of these patients, v) to estimate the effect of the intervention, both in the muscle strength and in post-intervention CPET, biochemical and anthropometric parameters, v) to estimate the effect of the intervention in the quality of life, anxiety, depression, and adherence to the Mediterranean diet.

DETAILED DESCRIPTION:
Methodology: our project is a quantitative study. Patients belonging to the integrated health area of the provinces Cuenca, Toledo, and Albacete will be included. The quantitative study will be a pre-post clinical trial in which at least 80 patients of both genders will be analyzed; who have suffered a coronary event in recent months.

Patients will receive a physical exercise intervention within a cardiac rehabilitation program, lasting 2 months, 3 days per week. The intervention consists of a first part of warm up the large muscle groups, accompanied by breathing exercises (10-15 minutes), followed by a part of strength and muscular resistance training exercises (upper and lower limbs and abdominal muscles), through an exercise table with weights of different weights, depending on the patient's 1RM (maximum repetition), elastic bands of different resistances and weights (15 minutes). Depending on the pathology, a series of special considerations will be taken into account regarding progressive loading (with weights) and resistance, degrees of joint mobility of the upper limbs.

The design of the strength and muscular resistance exercises will be planned taking into account heart rate (HR), cardiovascular pathology, physical capacity of the patient, hemodynamic response at rest, during exercise and after recovery from it, as well as the perception effort and pharmacological action.

Following the recommendations made by the existing literature, we will work the upper limb muscles with a load of 30-40% of the 1RM, with 50-60% of the 1RM being the workload prescribed for lower limb training. Next, we would move on to the aerobic exercise part (continuous and interval), using a treadmill or cycle ergometer, depending on the pathology and the individual characteristics of each patient. The objective we set for ourselves is to increase the duration and intensity progressively until we reach after 45 minutes, after a few weeks. The program would end with a cool-down phase or return to calm.

Study design: This project will have a quantitative design, specifically a pre-post clinical trial.

Patients aged between 20-80 with cardiovascular pathology meeting the inclusion criteria who will be referred from outpatient clinics, hospitalization or primary care and belonging to the provinces of Cuenca, Toledo, and Albacete will be included.

The participants under study will be recruited through their primary care doctor, or cardiologists from the provinces assigned to this project.

The study will be carried out at the "Virgen de la Luz Hospital", in Cuenca, among patients with cardiac pathology described in the inclusion criteria, who will be included in a cardiac rehabilitation program. The variables collected before and after the intervention will be analyzed and studied to assess the adherence of the program and the medium-long term objectives.

The recruitment of participants will be carried out throughout the entire project.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 20 and 80 years
2. Having suffered an acute event or presenting chronic cardiovascular pathology with a decrease/limitation of their functional capacity
3. Residing in the provinces of Cuenca, Toledo, or Albacete
4. Desire to participate voluntarily and acceptance of the conditions

Exclusion Criteria:

1. Have some physical or mental pathology that prevents their participation
2. Inability to adhere to the full program as reported in the initial consultation
3. Being outside the age criteria defined above

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen uptake | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in cardiorespiratory fitness | Baseline and at the end of the 8weeks intervention
  6 minutes walking test (6MWT)

SECONDARY OUTCOMES:
Change in blood pressure | Baseline and at the end of the 8weeks intervention
  Measured before and after the intervention with the Omron M7 Intelli blood pressure monitor
Change in basal heart rate | Baseline and at the end of the 8weeks intervention
  Measured before and after the intervention after CPET with the Omron M7 Intelli blood pressure monitor.
Change in Maximum heart rate: | Baseline and at the end of the 8weeks intervention
  Measured before and after the intervention after CPET with the Omron M7 Intelli blood pressure monitor
Change in oxygen consumption efficiency slope (OUES) | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in Respiratory gas exchange ratio (RER) | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in Ventilatory thresholds (VT1 -VT2) | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in Heart rate at ventilatory thresholds | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in ventilatory equivalents | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in partial pressures | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in oxygen pulse | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in ventilation (VE) | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in respiratory reserve (BR) | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in muscle efficiency | Baseline and at the end of the 8weeks intervention
  Cardiopulmonary exercise test (CPET)
Change in forced vital capacity (FVC) | Baseline and at the end of the 8weeks intervention
  Using spirometry
Change in forced expired volume in 1 second (FEV1) | Baseline and at the end of the 8weeks intervention
  Using spirometry
Changes in FEV1/FVC | Baseline and at the end of the 8weeks intervention
  Using spirometry
Changes in Maximum Flow 75 (MEF75)(Maximum Flow at 75% of Forced Vital Capacity) | Baseline and at the end of the 8weeks intervention
  Using spirometry
Changes in Maximum Flow 50 (MEF50) (Maximum Flow at 50% of Forced Vital Capacity) | Baseline and at the end of the 8weeks intervention
  Using spirometry
Changes in Maximum Flow 25 (MEF25) (Maximum Flow at 25% of Forced Vital Capacity) | Baseline and at the end of the 8weeks intervention
  Using spirometry
Changes in Peak expiratory flow (PEF) | Baseline and at the end of the 8weeks intervention
  Using spirometry
Changes in tidal volume (VC) | Baseline and at the end of the 8weeks intervention
  Using spirometry
Change in Weight | Baseline and at the end of the 8weeks intervention
  the mean of two measurements (using a OmronBF511 bioimpedance scale) with the participant barefoot and lightly clothed.
Change in Body mass index (BMI) | Baseline and at the end of the 8weeks intervention
  as weight (kg)/height2 (m2)
Change in Waist circumference | Baseline and at the end of the 8weeks intervention
  the mean of three measurements using a flexible tape measure at the midpoint between the last rib and the iliac crest at the end of a normal exhalation.
Change in Hip circumference | Baseline and at the end of the 8weeks intervention
  the mean of three measurements using a flexible tape measure between one and another greater trochanter.
Change in waist hip index | Baseline and at the end of the 8weeks intervention
  as waist circumference (cm)/ hip circumference (cm).
Change in Body fat percentage | Baseline and at the end of the 8weeks intervention
  the mean of two measurements using a OnromBF511 bioimpedance scale.
Change in HbA1c | Baseline and at the end of the 8weeks intervention
  Measured by blood test.
Change in total cholesterol | Baseline and at the end of the 8weeks intervention
  Measured by blood test.
Change in LDL-c cholesterol | Baseline and at the end of the 8weeks intervention
  Measured by blood test.
Change in HDL-c cholesterol | Baseline and at the end of the 8weeks intervention
  Measured by blood test.
Change in triglycerides | Baseline and at the end of the 8weeks intervention
  Measured by blood test.
Change in one repetition maximum (1RM) | Baseline and at the end of the 8weeks intervention
  Measured indirectly by Brzycki´s formula.
Change in handgrip in right arm | Baseline and at the end of the 8weeks intervention
  Measured by CAMRY digital dynamometer.
Change in handgrip in left arm | Baseline and at the end of the 8weeks intervention
  Measured by Camry digital dynamometer.
Change in maximum respiratory pressures | Baseline and at the end of the 8weeks intervention
  Measured by MicroMedical-Carefusion MicroRPM model.
Change in Health-related quality of life | Baseline and at the end of the 8weeks intervention
  36-Item Short Form Survey (SF-36)
Change in Depression and anxiety. | Baseline and at the end of the 8weeks intervention
  Hospital Anxiety and Depression Scale (HADS)
Change in adherence to the Mediterranean diet | Baseline and at the end of the 8weeks intervention
  Predimed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Priego-Jiménez, MsC, Principal Investigator — Hospital Virgen de la Luz; Laura Núñez-Martínez, MsC, Principal Investigator — Hospital Virgen de la Luz
Locations (1):
- Hospital Virgen de la Luz, Cuenca, Cuenca, Spain